CLINICAL TRIAL: NCT05484726
Title: Maternal Role in Sensory-motor Stimulation for Oral Feed Establishment in Preterm Neonates: MSMS Trial
Brief Title: Maternal Role in Oral Feed Establishment in Preterm Neonates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fatima Memorial Hospital (Other)
Responsible Party: Principal Investigator, Rafia Gul, Assistant Professor, Fatima Memorial Hospital
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Supportive Care
Other Study IDs: FMH-07-2021-IRB-929-M
Record Dates: First submitted 2022-07-30; First posted 2022-08-02 (Actual); Results first posted 2024-12-02 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-10

CONDITIONS: Preterm Birth; Tube Feeding; Swallowing Disorder; Maternal Care Patterns
Keywords: Prematurity; sensory-motor stimulation; oral feed establishment; feeding intervention
MeSH Terms: conditions — Premature Birth; Deglutition Disorders

STUDY DESIGN:
Intervention Model Description: 1. Maternal involvement in perioral sensory-motor stimulation be in three stages
     1. Observer status
     2. Performing under supervision
     3. Independent
  2. Intervention period: 5 days as
     1. Training phase (T): T1 and T2 (for mothers by the nurse)
     2. Direct feeding phase (D): F1, 2, and 3 (oral feed shall be offered to neonate)
  3. Stimulation for 7 minutes and 15 minutes before feeding twice a day at 1100 and 1700 hrs.
  4. Two groups
     1. Intervention group (GI): by mothers
     2. Control group (G II): by staff nurses
Who Masked: Care Provider
Masking Description: The mothers, medical staff involved in general care, nursing staff involved in the intervention, and doctors conducting the assessment of oral feeding skills (OFS) were all blinded to allocation. The nursing staff was informed at the time of intervention that participating infants would receive either sensory motor stimulation or sham oral stimulation depending on group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Group 1) (Experimental): * Maternal involvement shall be in three stages for the intervention group as
    * Observer status
    * Performing under supervision
    * Independent
  * Study groups for sensory motor stimulation (5 minutes) + pacifier (2 minutes)
  Intervention group (Group I): by mothers
  1. T1: Nurses performing all steps while mother observer status
  2. T2: Nurses perform all steps in front of the mother and a pacifier will be offered by the mother
  3. D1: Mother performs all steps and oral milk shall be offered by the nurse while the mother observes.
  4. D2: Mother performing all steps and offering oral milk while the nurse is supervising
  5. D3: Mother performing all steps independently
  Interventions: Other: perioral sensory motor stimulation
- Control group (Group 2) (Sham Comparator): All steps will be the same as the intervention group and shall be performed by staff nurses
  Interventions: Other: perioral sensory motor stimulation

INTERVENTIONS:
Other: perioral sensory motor stimulation — Step 1 - 6 over 5 minutes
  1 With the help of the index finger, on the external surface of the cheek, make a circle starting from the angle of the mouth towards the ear then back 7x each cheek
  2 While holding both sides of the cheek with help of the thumb and index finger repeat step 1 7x each cheek
  3 Move index finger from one corner to opposite one over both lips separately 7x each lip
  4 Gentle massage and compress the gums from center to back of mouth 7x each half of the gum
  5 Move the finger from front to back on the hard palate while applying gentle pressure 7x
  6 Displace the center of the tongue with gentle pressure 7x
  7 Offer pacifier at the end 2 minutes
  Note: 7x means 7 times

SUMMARY:
Hypothesis

Preterm babies who receive sensory motor stimulation from their mothers as compared to trained nurses will

1. Start taking oral feed at the same time as compared to control group
2. Take the same amount of milk at the commencement of oral feeding
3. Take milk with equal efficiency
4. Not face more adverse effects

DETAILED DESCRIPTION:
Aim To determine the maternal role in sensory-motor stimulation for oral feed establishment in preterm neonates Objective

1. Determine the effect of sensory-motor stimulation offered by the mother on the onset of oral feeding
2. Efficiency of mother-mediated stimulation techniques on oral feeding as compared to trained nurses
3. Study maternal role in the establishment of oral feed Hypothesis Preterm babies who receive sensory motor stimulation from their mothers as compared to trained nurses will

1. Start taking oral feed at the same time frame as compared to the control group 2. Take the very same amount of milk at the commencement of oral feeding 3. Take milk with equal efficiency 4. There is no extra burden of adverse effects

Data Collection All on going and related trials for this intervention shall be registered in the ClinicalTrials.gov. Study shall be conducted after ethical approval from IRB. All participants shall be enrolled after written informed consent from mothers after approval from attending neonatologist (annexure 2). All relevant maternal and neonatal data shall be collected on a specially designed proforma (annexure 3) with following details

1. Part 1: Maternal demographic and clinical data (age, parity, educational qualification, residence, previous preterm baby, job status, diabetes, hypertensive disorders, chronic ailment, multifetal gestation
2. Part 2: Neonatal demographic data (gender, gestation age, birth weight, growth centiles, diagnosis, APGAR score, noninvasive (NIV) and invasive ventilation with duration, caffeine, days taken for establishment of gavage feeding, age, and weight at commencement of intervention, any other complication during study)
3. Part 3: Neonatal feeding physiological measurements (SpO2, respiratory rate, heart rate before and after feeding, daily weight gain, type of milk offered)
4. Part 4: Oral feeding skill (OFS) assessment adapted from the model presented by Lau and Smith (p). All parameters shall be recorded twice a day for D1, D2, and D3 separately. It includes

   * Total volume prescribed (ml)
   * Total volume has taken during feeding (ml)
   * Volume has taken during the first 5 min of feeding (ml)
   * Duration of oral feeding (min)
   * Overall transfer (OT %) volume taken/total volume prescribed
   * Proficiency(PRO%) volume taken during the first 5 min/total volume prescribed
   * Rate of transfer (RT) ml/min
   * SSB (Suck Swallow Breaths) coordination
   * Adverse events (cough, fatigue)
   * According to this oral feeding ability can be classified into four levels depending upon the level of maturity in ascending order as follows:

     * Level 1: PRO < 30% and RT < 1.5 ml/min
     * Level 2: PRO < 30% and RT ≥ 1.5 ml/min
     * Level 3: PRO ≥ 30% and RT < 1.5 ml/min
     * Level 4: PRO ≥ 30% and RT ≥ 1.5 ml/min

ELIGIBILITY:
Inclusion Criteria:

* All preterm of gestation age 28 to 34weeks
* Haemodynamically stable
* Established full Gavage feed
* No respiratory distress
* No need for respiratory support except LFNC
* Do not receive any kind of analgesics

Exclusion Criteria:

* Syndromic babies /genetic disorders
* Haemodynamically unstable babies including IVH (grade III & IV), hemodynamically significant PDA on treatment, NEC(stage III)
* Major malformations
* Cleft lip and palate
* Anemia requiring blood transfusion

Ages: 30 Weeks to 34 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 130 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-09-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rafia Gul, FCPS (Neo), Principal Investigator — Fatima Memorial Hospital
Locations (1):
- Rafia Gul, Lahore, Shadman, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
After approval from the publishing journal once the study has been completed
Supporting Information: Study Protocol, SAP
Time Frame: 1 year after the study's publication for 3 months
Access Criteria: on request to corresponding author

REFERENCES:
- [Background] da Rosa Pereira K, Levy DS, Procianoy RS, Silveira RC. Impact of a pre-feeding oral stimulation program on first feed attempt in preterm infants: Double-blind controlled clinical trial. PLoS One. 2020 Sep 9;15(9):e0237915. doi: 10.1371/journal.pone.0237915. eCollection 2020. PMID 32903261
- [Background] Murthy SV, Funderburk A, Abraham S, Epstein M, DiPalma J, Aghai ZH. Nasogastric Feeding Tubes May Not Contribute to Gastroesophageal Reflux in Preterm Infants. Am J Perinatol. 2018 Jun;35(7):643-647. doi: 10.1055/s-0037-1608875. Epub 2017 Nov 30. PMID 29190845
- [Background] Rogers SP, Hicks PD, Hamzo M, Veit LE, Abrams SA. Continuous feedings of fortified human milk lead to nutrient losses of fat, calcium and phosphorous. Nutrients. 2010 Mar;2(3):230-40. doi: 10.3390/nu2030240. Epub 2010 Feb 26. PMID 22254018
- [Background] Viswanathan S, Jadcherla S. Transitioning from gavage to full oral feeds in premature infants: When should we discontinue the nasogastric tube? J Perinatol. 2019 Sep;39(9):1257-1262. doi: 10.1038/s41372-019-0446-2. Epub 2019 Jul 31. PMID 31366911
- [Background] Greene Z, O'Donnell CP, Walshe M. Oral stimulation for promoting oral feeding in preterm infants. Cochrane Database Syst Rev. 2016 Sep 20;9(9):CD009720. doi: 10.1002/14651858.CD009720.pub2. PMID 27644167
- [Background] 6. Maltese A, Gallai B, Marotta R, Lavano F, Lavano S, Tripi G. The synactive theory of development: the keyword for neurodevelopmental disorders. Acta Medica Mediterranea, 2017, 33: 1257-63
- [Background] Song D, Jegatheesan P, Nafday S, Ahmad KA, Nedrelow J, Wearden M, Nemerofsky S, Pooley S, Thompson D, Vail D, Cornejo T, Cohen Z, Govindaswami B. Patterned frequency-modulated oral stimulation in preterm infants: A multicenter randomized controlled trial. PLoS One. 2019 Feb 28;14(2):e0212675. doi: 10.1371/journal.pone.0212675. eCollection 2019. PMID 30817764
- [Background] Bertoncelli N, Cuomo G, Cattani S, Mazzi C, Pugliese M, Coccolini E, Zagni P, Mordini B, Ferrari F. Oral feeding competences of healthy preterm infants: a review. Int J Pediatr. 2012;2012:896257. doi: 10.1155/2012/896257. Epub 2012 May 17. PMID 22675368
- [Background] Simpson C, Schanler RJ, Lau C. Early introduction of oral feeding in preterm infants. Pediatrics. 2002 Sep;110(3):517-22. doi: 10.1542/peds.110.3.517. PMID 12205253
- [Background] Lau C, Sheena HR, Shulman RJ, Schanler RJ. Oral feeding in low birth weight infants. J Pediatr. 1997 Apr;130(4):561-9. doi: 10.1016/s0022-3476(97)70240-3. PMID 9108854
- [Background] Sarin E, Maria A. Acceptability of a family-centered newborn care model among providers and receivers of care in a Public Health Setting: a qualitative study from India. BMC Health Serv Res. 2019 Mar 21;19(1):184. doi: 10.1186/s12913-019-4017-1. PMID 30898170
- [Background] 13. Fonseca SA, Silveira AO, Franzoi MAH, Motta E. Family centered-care at the neonatal intensive care unit (NICU): nurses' experiences. Enfermería: Cuidados Humanizados. 2020; 9(2): 170-190
- [Background] Ghomi H, Yadegari F, Soleimani F, Knoll BL, Noroozi M, Mazouri A. The effects of premature infant oral motor intervention (PIOMI) on oral feeding of preterm infants: A randomized clinical trial. Int J Pediatr Otorhinolaryngol. 2019 May;120:202-209. doi: 10.1016/j.ijporl.2019.02.005. Epub 2019 Feb 5. PMID 30851536
- [Background] Fucile S, Gisel EG, McFarland DH, Lau C. Oral and non-oral sensorimotor interventions enhance oral feeding performance in preterm infants. Dev Med Child Neurol. 2011 Sep;53(9):829-835. doi: 10.1111/j.1469-8749.2011.04023.x. Epub 2011 Jun 27. PMID 21707601
- [Background] Lau C, Smith EO. A novel approach to assess oral feeding skills of preterm infants. Neonatology. 2011;100(1):64-70. doi: 10.1159/000321987. Epub 2011 Jan 5. PMID 21212698
- [Background] Majoli M, De Angelis LC, Panella M, Calevo MG, Serveli S, Knoll BL, Ramenghi LA. Parent-Administered Oral Stimulation in Preterm Infants: A Randomized, Controlled, Open-Label Pilot Study. Am J Perinatol. 2023 Jun;40(8):845-850. doi: 10.1055/s-0041-1731452. Epub 2021 Jun 28. PMID 34182577

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study period spans 16 months (March 2022 - July 2023), in the department of Neonatology, Fatima Memorial Hospital, Lahore. All preterm of gestation age 28 to 34 weeks, admitted to NICU during the study period after seeking consent from parents or guardians were enrolled. All neonates having major anomalies incompatible with life, cleft lip and palate, genetic disorders, IVH (grade III & IV), HsPDA, hemodynamic instability, NEC (stage II & III) or anemia requiring transfusion were excluded.
Pre-assignment Details: Out of 142 eligible neonates, study was started with 130 as 65 in each group. Twelve neonates were excluded as 2 mothers experienced serious postnatal complications, 1 instance of parental refusal after initial participation, 1 case with incomplete data, and 8 others.
  Out of 65 neonates in each group, in 49 from intervention group and 48 from control group, sensory motor stimulation could be performed per protocol as 33 total neonates were excluded and details have been mentioned in table.
Groups:
- Intervention Group (Group 1): * Maternal involvement was done in three stages for the intervention group as
    o Observer status
    * Performing under supervision
    * Independent
  * Study groups for sensory motor stimulation (5 minutes) + pacifier (2 minutes)
  Intervention group (Group I): by mothers
  1. T1: Nurses performed all steps while mother observer status
  2. T2: Nurses performed all steps in front of the mother and a pacifier was offered by the mother
  3. D1: Mother performed all steps and oral milk was offered by the nurse while the mother observed.
  4. D2: Mother performed all steps and offering oral milk under nurse supervision
  5. D3: Mother performed all steps independently
  perioral sensory motor stimulation: Step 1 - 6 over 5 minutes
  1 With the help of the index finger, on the external surface of the cheek, make a circle starting from the angle of the mouth towards the ear then back 7x each cheek
  2 While holding both sides of the cheek with help of the thumb and index finger repeat step 1 7x each cheek
  3 Move index finger from one corner to opposite one over both lips separately 7x each lip
  4 Gentle massage and compress the gums from center to back of mouth 7x each half of the gum
  5 Move the finger from front to back on the hard palate while applying gentle pressure 7x
  6 Displace the center of the tongue with gentle pressure 7x
  7 Offer pacifier at the end 2 minutes
  Note: 7x means 7 times
- Control Group (Group 2): All steps were the same as the intervention group and were performed by staff nurses
  perioral sensory motor stimulation: Step 1 - 6 over 5 minutes
  1 With the help of the index finger, on the external surface of the cheek, make a circle starting from the angle of the mouth towards the ear then back 7x each cheek
  2 While holding both sides of the cheek with help of the thumb and index finger repeat step 1 7x each cheek
  3 Move index finger from one corner to opposite one over both lips separately 7x each lip
  4 Gentle massage and compress the gums from center to back of mouth 7x each half of the gum
  5 Move the finger from front to back on the hard palate while applying gentle pressure 7x
  6 Displace the center of the tongue with gentle pressure 7x
  7 Offer pacifier at the end 2 minutes
  Note: 7x means 7 times
Period: Overall Study
Arm/Group | Intervention Group (Group 1) | Control Group (Group 2)
Started | 65 | 65
Execution of Sensory Motor Stimulation (neonates were stable to start with oromotor stimulation followed by feeding.) | 54 | 53
Completed | 49 | 48
Not Completed | 16 | 17
Not completed — Protocol Violation | 3 | 3
Not completed — failure to establish gavage feed by 2 weeks of chronological age | 4 | 2
Not completed — HsPDA requiring antifailure therapy | 1 | 2
Not completed — continued need of mechanical ventilation | 2 | 3
Not completed — Withdrawal by Subject | 2 | 3
Not completed — IVH (G III & IV) | 2 | 1
Not completed — NEC (stage II & III) | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Intervention Group (Group 1): Maternal involvement was done in three stages for the intervention group as
  * Observer status
  * Performing under supervision
  * Independent
    * Study groups for sensory motor stimulation (5 minutes) + pacifier (2 minutes) Intervention group (Group I): by mothers
      1. T1: Nurses performed all steps while mother observer status
      2. T2: Nurses performed all steps in front of the mother and a pacifier was offered by the mother
      3. D1: Mother performed all steps and oral milk was offered by the nurse while the mother observed.
      4. D2: Mother performed all steps and offering oral milk under nurse supervision
      5. D3: Mother performed all steps independently perioral sensory motor stimulation: Step 1 - 6 over 5 minutes
      <!-- -->
      1. With the help of the index finger, on the external surface of the cheek, make a circle starting from the angle of the mouth towards the ear then back 7x each cheek
      2. While holding both sides of the cheek with help of the thumb and index finger repeat step 1 7x each cheek
      3. Move index finger from one corner to opposite one over both lips separately 7x each lip
      4. Gentle massage and compress the gums from center to back of mouth 7x each half of the gum
      5. Move the finger from front to back on the hard palate while applying gentle pressure 7x
      6. Displace the center of the tongue with gentle pressure 7x
      7. Offer pacifier at the end 2 minutes Note: 7x means 7 times
- Total: Total of all reporting groups
Arm/Group | Intervention Group (Group 1) | Control Group (Group 2) | Total
Number analyzed (Participants) | 49 | 48 | 97
Age, Continuous [Median (Inter-Quartile Range); unit: years] — maternal age at time of delivery measured as years
  years | 29 [26 to 32] | 30 [26.5 to 33] | 29.5 [26.3 to 32.5]
Sex/Gender, Customized [Count of Participants; unit: Participants] — all mothers were female
  Participants | 49 | 48 | 97
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Maternal education [Count of Participants; unit: Participants]
  Uneducated | 2 | 2 | 4
  Primary | 11 | 10 | 21
  Secondary | 15 | 20 | 35
  Higher | 21 | 16 | 37
mothers with previous preterm neonates [Count of Participants; unit: Participants] | 42 | 38 | 80
Maternal Job status [Count of Participants; unit: Participants]
  home maker | 29 | 31 | 60
  job doing | 20 | 17 | 37
hypertensive disorder of pregnancy [Count of Participants; unit: Participants] — maternal record of blood pressure during pregnancy was used to diagnose pregnancy induced hypertension
  Participants | 29 | 32 | 61
Gestational diabetes mellitus [Count of Participants; unit: Participants] — diabetes mellitus was diagnosed in pregnancy by measuring blood sugar level by 20 weeks of gestation or later
  Participants | 17 | 17 | 34
anemia of pregnancy [Count of Participants; unit: Participants] — Maternal hemoglobin of < 10 mg/dl was labelled as anemia of pregnancy
  Participants | 25 | 21 | 46
Gravidity [Count of Participants; unit: Participants]
  Primigravida (PG) | 20 | 26 | 46
  2 - 3 | 22 | 15 | 37
  4 or more | 7 | 7 | 14
neonatal gender (male) [Count of Participants; unit: Participants] | 27 | 22 | 49
Gestation age at delivery [Median (Inter-Quartile Range); unit: weeks] | 30 [29 to 32] | 31 [29.3 to 32] | 30.5 [29.2 to 32]
Mode of delivery (SVD) [Count of Participants; unit: Participants] | 26 | 29 | 55
Birth weight [Median (Inter-Quartile Range); unit: Kg] | 1.29 [1.20 to 1.52] | 1.34 [1.15 to 1.67] | 1.31 [1.18 to 1.60]
Weight for gestational age [Count of Participants; unit: Participants] — neonatal weight was plotted for gestation age on gender specific growth chart to determine weight for gestation age
  Participants
    Appropriate for gestation age (AGA) | 27 | 30 | 57
    Small for gestation age (SGA) | 16 | 15 | 31
    Large for gestation age (LGA) | 6 | 3 | 9
Place of birth (Inborn) [Count of Participants; unit: Participants] — In born were all those neonates who were born in our own hospital
  Participants | 30 | 33 | 63
Required Invasive mechanical ventilation (IMV) [Count of Participants; unit: Participants] | 26 | 30 | 56
Duration of IMV [Median (Inter-Quartile Range); unit: days] — Population: the number of neonates receiving IMV
  days
    number analyzed (Participants) | 26 | 30 | 56
    (all) | 1 [0 to 4] | 2 [0 to 5] | 1.5 [0 to 4.5]
Required non invasive ventilation (NIV) [Count of Participants; unit: Participants] — all neonates had respiratory failure and were spontaneously breathing require non invasive ventilation (NIV)
  Participants | 45 | 48 | 93
Duration of non invasive ventilation (NIV) [Median (Inter-Quartile Range); unit: days] — for only those neonates who received non invasive ventilation Population: Only those neonates who received non invasive ventilation (NIV)
  days
    number analyzed (Participants) | 45 | 48 | 93
    (all) | 3 [1 to 7] | 4 [2 to 6.75] | 3.5 [1.5 to 6.9]
Required low flow nasal cannula therapy (LFNC) [Count of Participants; unit: Participants] — All neonates with type 1 respiratory failure requiring oxygen only to maintain their oxygen saturation
  Participants | 47 | 43 | 90
Duration of LFNC [Median (Inter-Quartile Range); unit: days] — only those neonates who required low flow nasal cannula therapy (LFNC) Population: Only those neonates were analysed who required LFNC
  days
    number analyzed (Participants) | 47 | 43 | 90
    (all) | 4 [2 to 5] | 3.5 [2 to 5] | 3.75 [2 to 5]
Apnea [Count of Participants; unit: Participants] — Apnea was diagnosed on basis of breath holding spells for > 20 second with or without bradycardia
  Participants | 18 | 20 | 38
Respiratory distress syndrome (RDS) [Count of Participants; unit: Participants] — Respiratory distress syndrome (RDS) was diagnosed on clinical and radiological features of reticulo-nodular shadowing
  Participants | 25 | 25 | 50
Caffeine [Count of Participants; unit: Participants] — Use of prophylactic caffeine therapy as yes or now. It was given to all neonates < 32 weeks of gestation age as started on first day of life to avoid apnea of prematurity.
  Participants | 28 | 28 | 56
Hemodynamically significant patent ductus arteriosus (HsPDA) [Count of Participants; unit: Participants] | 17 | 20 | 37
Necrotizing enterocolitis (NEC) [Count of Participants; unit: Participants] | 9 | 12 | 21
Feeding intolerence [Count of Participants; unit: Participants] | 20 | 25 | 45
Sepsis [Count of Participants; unit: Participants] | 43 | 41 | 84
Seizures [Count of Participants; unit: Participants] | 7 | 5 | 12
Post menstural age (PMA) at enrollment [Median (Inter-Quartile Range); unit: weeks] | 32 [31 to 33] | 32 [31 to 33] | 32 [31 to 33]
Chronological age (ChA) at enrollment [Median (Inter-Quartile Range); unit: days] | 13 [6 to 14] | 9 [7 to 16] | 11 [6.5 to 11]
Time to full gavage feed [Median (Inter-Quartile Range); unit: days] | 7 [5.5 to 13.5] | 7 [6 to 14] | 7 [5.7 to 13.7]
Discharge weight [Median (Inter-Quartile Range); unit: Kg] | 1.48 [1.42 to 1.66] | 1.48 [1.43 to 1.75] | 1.48 [1.42 to 1.7]
Weight at enrollment [Median (Inter-Quartile Range); unit: Kg] | 1.35 [1.25 to 1.54] | 1.35 [1.21 to 1.60] | 1.35 [1.21 to 1.57]
Duration of stay in NICU [Median (Inter-Quartile Range); unit: days] | 21 [15 to 29.5] | 30 [16 to 30.75] | 25.5 [15.5 to 30.1]

OUTCOME MEASURES:

1. Primary Outcome: Transition Time to Full Oral Feeding
Description: Time interval between commencement of perioral sensory stimulation on D1 to establishment of full oral feed in both groups. It was done daily till 14th day of perioral sensory motor stimulation. Transition time to full oral feeding was the day at which baby was able to take oral feed of volume of 120-140ml/kg/day.
Time Frame: Expected time of oral feed establishment
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Intervention Group (Group 1) | Control Group (Group 2)
Number analyzed (Participants) | 49 | 48
days | 10 [7 to 13] | 9 [7 to 13]

2. Primary Outcome: Improvement (Change) in Efficiency in Oral Feed Establishment
Description: According to this efficiency in oral feed establishment in terms of amount and time is determined for the intervention group vs the control group.
  It can be classified into four levels depending upon the level of maturity in ascending order as follows:
  * Level 1: PRO < 30% and RT < 1.5 ml/min
  * Level 2: PRO < 30% and RT ≥ 1.5 ml/min
  * Level 3: PRO ≥ 30% and RT < 1.5 ml/min
  * Level 4: PRO ≥ 30% and RT ≥ 1.5 ml/min For all neonates, efficacy was measured at 11.00 am and 5.00 pm following sensory motor stimulation for both groups till achievement of full oral feed.
Time Frame: For record purpose in this study results, efficacy level was noted as L4 on the following days D1, D2, D3, D5, D7 and D14
Population: neonates were assessed for efficacy of level 4 (L4) on D1, D2,D3,D5,D7 and D14
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group (Group 2) | Intervention Group (Group 1)
Number analyzed (Participants) | 48 | 49
Participants
  L4 efficacy by D1-3 | 0 | 0
  L4 efficacy by D5 | 9 | 12
  L4 efficacy by D7 | 15 | 16
  L4 efficacy by D14 | 36 | 35

3. Primary Outcome: •Adverse Outcome Monitoring
Description: monitor for any adverse events like cough, breath holding, chocking, aspiration, tachycardia, and or bradycardia with
  1. stimulation
  2. feed Adverse outcome monitoring as non-life threatening adverse events including cough, tachycardia HR 180-200/min, bradycardia HR120 - 100/min, , tachypnea RR 60 - 70/min while maintaining SpO2 of >90% at room air
Time Frame: Adverse events were noted on D1, D2,D3,D5,D7 and D14
Population: All neonates were monitored for adverse outcome. This monitoring was done as non-life threatening adverse events including cough, tachycardia HR 180-200/min, bradycardia HR120 - 100/min, , tachypnea RR 60 - 70/min while maintaining SpO2 of >90% at room air
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group (Group 2) | Intervention Group (Group 1)
Number analyzed (Participants) | 48 | 49
Participants
  Adverse events D1 | 31 | 36
  Adverse events D2 | 14 | 14
  Adverse events D3 | 12 | 12
  Averse events D5 | 0 | 2
  Adverse events D7 & 14 | 0 | 0

4. Secondary Outcome: • Total Volume Taken During Each Feeding
Description: It is the measure of how much feed has been taken orally out of total feed prescribed for each feeding
Time Frame: It was noted on D1, D2, D3, D5, D7 and D14
Measure: Median (Inter-Quartile Range); unit: ml
Arm/Group | Control Group (Group 2) | Intervention Group (Group 1)
Number analyzed (Participants) | 48 | 49
ml
  Oral feed volume/feed on D1 | 2 [2 to 7] | 2 [2 to 7]
  Oral feed volume/feed on D2 | 3 [2 to 7] | 5 [2 to 9]
  Oral feed volume/feed on D3 | 4 [3 to 10] | 7 [3 to 11]
  Oral feed volume/feed on D5 | 6.5 [5 to 15] | 8 [5 to 15]
  Oral feed volume/feed on D7 | 7.5 [7 to 20] | 9 [7 to 18]
  Oral feed volume/feed on D14 | 15.5 [14 to 22] | 15.5 [13 to 20.5]

5. Secondary Outcome: • Volume Taken During the First 5 Min of Feeding (ml) VT5
Description: during each feed taken orally by neonate VT5 is the amount of feed was taken by neonate during first 5 minutes
Time Frame: Volume taken during the first 5 min of feeding (ml) VT5 was measured on D1, D2, D3, D5, D7 and D14
Measure: Median (Inter-Quartile Range); unit: ml
Arm/Group | Control Group (Group 2) | Intervention Group (Group 1)
Number analyzed (Participants) | 48 | 49
ml
  VT5 on D1 | 2 [1.25 to 4] | 2 [1 to 4.5]
  VT5 on D2 | 3 [2 to 5] | 3 [2 to 6]
  VT5 on D3 | 3 [2 to 7] | 3 [2 to 7]
  VT5 on D5 | 5 [4 to 8] | 5 [4 to 9]
  VT5 on D7 | 7 [6 to 10] | 7 [5.5 to 11]
  VT5 on D14 | 10 [9 to 10] | 10 [9 to 12.5]

6. Secondary Outcome: •Rate of Transfer (RT) ml/Min
Description: RT is the time taken by neonate to finish oral feed
Time Frame: RT was measured on D1, D2, D3, D5, D7 and D14
Measure: Median (Inter-Quartile Range); unit: ml/min
Arm/Group | Control Group (Group 2) | Intervention Group (Group 1)
Number analyzed (Participants) | 48 | 49
ml/min
  RT on D1 | 0.42 [0.28 to 0.70] | 0.42 [0.24 to 0.85]
  RT on D2 | 0.71 [0.70 to 1.0] | 0.70 [0.59 to 1.0]
  RT on D3 | 0.70 [0.4 to 1.0] | 0.70 [0.4 to 1.0]
  RT on D5 | 0.90 [0.50 to 1.2] | 0.83 [0.50 to 1.45]
  RT on D7 | 1.0 [0.67 to 1.7] | 1.0 [0.68 to 1.6]
  RT on D14 | 1.6 [1.1 to 2.1] | 1.6 [1.1 to 2.1]

7. Secondary Outcome: • Overall Transfer (OT Percent) Volume Taken/Total Volume Prescribed
Description: trend towards oral feed establishment and is measured as overall transfer of milk yo oral out of total amount prescribed
Time Frame: OT was measured on D1, D2, D3, D5, D7 and D14
Measure: Median (Inter-Quartile Range); unit: percentage of volume taken/total volume
Arm/Group | Control Group (Group 2) | Intervention Group (Group 1)
Number analyzed (Participants) | 48 | 49
percentage of volume taken/total volume
  OT on D1 | 21 [15.3 to 36] | 21 [15 to 36]
  OT on D2 | 35.7 [15 to 36] | 36 [15 to 44]
  OT on D3 | 43.8 [21 to 50] | 43.8 [21 to 55.5]
  OT on D5 | 48 [33 to 65] | 48 [33 to 65]
  OT on D7 | 56 [46 to 100] | 60 [46 to 73.5]
  OT on D14 | 95.5 [87.9 to 100] | 91 [87 to 100]

8. Secondary Outcome: • Proficiency(PRO Percent) Volume Taken During the First 5 Min/Total Volume Prescribed
Description: how much amount of milk is taken during first 5 minutes while administering oral feeding
Time Frame: PRO % was measured on D1, D2, D3, D5, D7 and D14
Measure: Median (Inter-Quartile Range); unit: percentage of volume taken during the fi
Arm/Group | Control Group (Group 2) | Intervention Group (Group 1)
Number analyzed (Participants) | 48 | 49
percentage of volume taken during the fi
  PRO on D1 | 16 [9.2 to 21] | 16 [7.8 to 24]
  PRO on D2 | 21 [15 to 27] | 21.6 [15 to 32.5]
  PRO on D3 | 19.5 [14 to 31] | 23 [14 to 37]
  PRO on D5 | 29 [24.5 to 39] | 30 [25 to 39]
  PRO on D7 | 39 [32 to 46] | 39 [33 to 49.5]
  PRO on D14 | 55.8 [46 to 56] | 56 [50 to 60]

9. Secondary Outcome: • Neonates Feeding With SSB Coordination
Description: number of neonates who are feeding well and showing coordinated pattern of suck swallow and breath (SSB)
Time Frame: It was measured on D1, D2, D3, D5, D7 and D14
Measure: Count of Participants; unit: Participants
Groups:
- Experimental Group (Group 1): Maternal involvement was done in three stages for the intervention group as
  * Observer status
  * Performing under supervision
  * Independent
    * Study groups for sensory motor stimulation (5 minutes) + pacifier (2 minutes) Intervention group (Group I): by mothers
      1. T1: Nurses performed all steps while mother observer status
      2. T2: Nurses performed all steps in front of the mother and a pacifier was offered by the mother
      3. D1: Mother performed all steps and oral milk was offered by the nurse while the mother observed.
      4. D2: Mother performed all steps and offering oral milk under nurse supervision
      5. D3: Mother performed all steps independently perioral sensory motor stimulation: Step 1 - 6 over 5 minutes
      <!-- -->
      1. With the help of the index finger, on the external surface of the cheek, make a circle starting from the angle of the mouth towards the ear then back 7x each cheek
      2. While holding both sides of the cheek with help of the thumb and index finger repeat step 1 7x each cheek
      3. Move index finger from one corner to opposite one over both lips separately 7x each lip
      4. Gentle massage and compress the gums from center to back of mouth 7x each half of the gum
      5. Move the finger from front to back on the hard palate while applying gentle pressure 7x
      6. Displace the center of the tongue with gentle pressure 7x
      7. Offer pacifier at the end 2 minutes Note: 7x means 7 times
Arm/Group | Control Group (Group 2) | Experimental Group (Group 1)
Number analyzed (Participants) | 48 | 49
Participants
  SSB on D1 | 23 | 22
  SSB on D2 | 27 | 33
  SSB on D3 | 32 | 33
  SSB on D5 | 37 | 40
  SSB on D7 | 36 | 39
  SSB on D14 | 48 | 49

10. Primary Outcome: •Adverse Events Monitoring
Description: as for outcome 3
Time Frame: Adverse events were noted on D1, D2,D3,D5,D7 and D14
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group (Group 2) | Intervention Group (Group 1)
Number analyzed (Participants) | 48 | 49
Participants
  Adverse events D1 | 31 | 36
  Adverse events D2 | 14 | 14
  Adverse events D3 | 12 | 12
  Averse events D5 | 0 | 2
  Adverse events D7 & 14 | 0 | 0

ADVERSE EVENTS:
Time Frame: For every neonate adverse events were monitored from first day (D1) of perioral sensory - motor stimulation to day of full oral feed establishment expected by Day 14
Description: Only those neonates were enrolled in study who were stable enough to tolerate the procedure of sensory motor stimulation and feeding.
Groups:
- Intervention Group (Group 1): * Maternal involvement shall be in three stages for the intervention group as
    o Observer status
    * Performing under supervision
    * Independent
  * Study groups for sensory motor stimulation (5 minutes) + pacifier (2 minutes)
  Intervention group (Group I): by mothers
  1. T1: Nurses performing all steps while mother observer status
  2. T2: Nurses perform all steps in front of the mother and a pacifier will be offered by the mother
  3. D1: Mother performs all steps and oral milk shall be offered by the nurse while the mother observes.
  4. D2: Mother performing all steps and offering oral milk while the nurse is supervising
  5. D3: Mother performing all steps independently
  perioral sensory motor stimulation: Step 1 - 6 over 5 minutes
  1 With the help of the index finger, on the external surface of the cheek, make a circle starting from the angle of the mouth towards the ear then back 7x each cheek
  2 While holding both sides of the cheek with help of the thumb and index finger repeat step 1 7x each cheek
  3 Move index finger from one corner to opposite one over both lips separately 7x each lip
  4 Gentle massage and compress the gums from center to back of mouth 7x each half of the gum
  5 Move the finger from front to back on the hard palate while applying gentle pressure 7x
  6 Displace the center of the tongue with gentle pressure 7x
  7 Offer pacifier at the end 2 minutes
  Note: 7x means 7 times
- Control Group (Group 2): All steps will be the same as the intervention group and shall be performed by staff nurses
  perioral sensory motor stimulation: Step 1 - 6 over 5 minutes
  1 With the help of the index finger, on the external surface of the cheek, make a circle starting from the angle of the mouth towards the ear then back 7x each cheek
  2 While holding both sides of the cheek with help of the thumb and index finger repeat step 1 7x each cheek
  3 Move index finger from one corner to opposite one over both lips separately 7x each lip
  4 Gentle massage and compress the gums from center to back of mouth 7x each half of the gum
  5 Move the finger from front to back on the hard palate while applying gentle pressure 7x
  6 Displace the center of the tongue with gentle pressure 7x
  7 Offer pacifier at the end 2 minutes
  Note: 7x means 7 times
Arm/Group | Intervention Group (Group 1) | Control Group (Group 2)
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/48
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/48
Other Adverse Events (participants affected / at risk) | 16/49 | 19/48
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Intervention Group (Group 1) (N=49) | Control Group (Group 2) (N=48)
Non-life threatening adverse events (Injury, poisoning and procedural complications) | 16 | 19 — cough, tachycardia HR 180-200/min, bradycardia HR120 - 100/min, , tachypnea RR 60 - 70/min while maintaining SpO2 of >90% at room air

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2024-04-21): https://cdn.clinicaltrials.gov/large-docs/26/NCT05484726/Prot_SAP_ICF_000.pdf